CLINICAL TRIAL: NCT03122795
Title: Sinonasal Microbiome Transplant as a Therapy for Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Snortransplantationsstudie1
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Patients and donors who meet the inclusion criteria will be recruited and inclueded and put through the study in a cumulative fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microbiome transplant (Experimental): The only arm of the study. Patients suffering from CRSsNP gets microbiome transplants from donors without any sinonasal health problems.
  Interventions: Procedure: Microbiome transplant

INTERVENTIONS:
Procedure: Microbiome transplant — A raw microbiome, collected from a donor without any sinonasal health problems, as a nasal lavage.

SUMMARY:
Chronic rhinosinusitis (CRS) is a disease associated with impaired quality of life and substantial societal costs. Though sometimes co-appearing with other conditions, such as asthma, allergy, and nasal polyps, many cases present without co-morbidities. Micro-biological diagnostic procedures are frequently undertaken, but the results are often inconclusive. Nevertheless, antibiotics are usually prescribed, but invariably with limited and temporary success. Accordingly, there is a need for new treatments for CRS.

Recent studies indicate that the sinuses are colonized by a commensal microbiome of bacteria and that damage to this natural microbiome, by pathogens or antibiotics, may cause an imbalance that may promote CRS. Therefore, treatments that restore the commensal microbiome may offer an alternative to current protocols. Arguably, as suggested by studies on patients with intestinal infections (next paragraph), one such possibility may be to transfer a "normal microbiome" to patients with CRS.

A disrupted microbiome is linked to intestinal clostridium difficile infections. Probiotic restitution therapy may be effective even in cases recalcitrant to antibiotic treatment. However, a key to effective probiotic restitution is selecting the bacteria that facilitate regrowth of normal microbiome. As an answer to this, researchers have chosen to simply transplant the entire microbiome from a healthy donor. In the case of clostridium difficile infection in the form of faecal transplants.

In this study, we will examine the possibility to treat patients with chronic rhinosinusitis without polyps (CRSsNP) with complete sinonasal microbiomes obtained from healthy donors. Our analysis will focus on symptoms and signs of disease as well as on nasal inflammatory and microbiological indices.

DETAILED DESCRIPTION:
Over the last few years the theory of a damaged microbiome as a cause or promoting factor behind chronic rhinosinusitis has gained increasing interest from the scientific community.

A number of studies aimed at investigating the microbiota of the nose and paranasal sinuses in health and disease has been published with very varying outcomes. Furthermore, other studies have been aimed at probiotic treatment of sinonasal disease either locally or through immunologic manipulation via the gastrointestinal microbiota.

A problem common to all these studies is that studies examining the normal nasal microbiota have identified a great amount of different bacterial species. It is as of today not known which individual species or combinations of species that promotes health.

The probiotic assemblages examined in previous studies have consisted of one or a combination of a few bacterial species.

Probiotic restitution therapy has been proven very effective for intestinal clostridium difficile infections. The restitution therapy has then consisted of transplantation of a complete microbiome from a healthy donor in the form of a faecal transplant.

In this study the investigators aim at recruiting patients suffering from chronic rhinosinusitis without polyps (CRSsNP) and healthy participants without any history sinonasal disease. The patients and the healthy participants will be examined for infectious diseases in a manner similar to other medical transplant procedures to minimize the risk for the recipients. The patients will then be treated with antibiotics to reduce the bacterial load of the nose and the paranasal sinuses. After the patient has finished the antibiotic treatment a microbiome transplant will be harvested from the healthy participant as a nasal lavage. The raw lavage fluid will then be used to transplant the microbiome to the patient. The procedure will be repeated for five consecutive days.

The outcome measures analysed will focus on subjective sinonasal health and symptoms of the patients but also include nasal inflammatory and microbiological indices.

ELIGIBILITY:
Inclusion criteria (patient)

* 2 nasal symptoms: 1 of which must be nasal obstruction or discoloured discharge.
* Sinusitis verified by endoscopy or CT-scan.
* Duration > 12 weeks.
* Previous surgery with patent ostia to the diseased sinuses.
* Signed informed consent to participate in the study.

Inclusion criteria (donor)

* No history of sinonasal or lower airway disease within the last 2 years other than the common cold.
* Accepted as a donor by the patient.
* Signed informed consent to participate in the study.

Exclusion criteria (patient)

* Nasal polyposis.
* Antibiotic treatment within the last 4 weeks.
* On-going or recent participation in another clinical trial.
* Any medication that may affect the results in an unpredictable manner.
* Immune deficiency.
* Allergy to amoxicillin or clavulanate potassium and clarithromycin.
* Pregnancy or breastfeeding.

Exclusion criteria (donor)

* Chronic rhinosinusitis.
* Acute rhinosinusitis within the last two years.
* Nasal polyposis.
* Asthma.
* Antibiotic treatment within the last 4 weeks.
* On-going or recent participation in another clinical trial.
* Clinical findings of sinonasal disease at the inclusion visit.
* Findings in the pre-study pathogen scan that makes the donor unsuitable.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
SNOT-22 | Day 1 to day 106
  Change of burden of disease as measured by the SNOT-22 (22 item sinonasal outcome test) questionnaire in patients

SECONDARY OUTCOMES:
Lund Kennedy endoscopy score | Day 1 to day 106
  Grading of burden of disease as measured using the Lund-Kennedy endoscopy score.
Subjective symptom score | Day 1 to 106.
  Subjective scoring of symptoms related to sinonasal, lower airway, intestinal and other
Inflammatory burden | Day 1 to day 106
  Amount of inflammatory mediators collected in nasal lavages.
Microflora | Day 1 to day 106
  Change in nasal microflora measured using both culture dependant and non culture dependant microbiological techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Mårtensson, MD, Principal Investigator — Region Skåne
Locations (1):
- Departement of ORL, Helsingborg, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will be presented at group level for personal integrity reasons.

REFERENCES:
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Background] Human Microbiome Project Consortium. Structure, function and diversity of the healthy human microbiome. Nature. 2012 Jun 13;486(7402):207-14. doi: 10.1038/nature11234. PMID 22699609
- [Background] Abreu NA, Nagalingam NA, Song Y, Roediger FC, Pletcher SD, Goldberg AN, Lynch SV. Sinus microbiome diversity depletion and Corynebacterium tuberculostearicum enrichment mediates rhinosinusitis. Sci Transl Med. 2012 Sep 12;4(151):151ra124. doi: 10.1126/scitranslmed.3003783. PMID 22972842
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Nagalingam NA, Cope EK, Lynch SV. Probiotic strategies for treatment of respiratory diseases. Trends Microbiol. 2013 Sep;21(9):485-92. doi: 10.1016/j.tim.2013.04.008. Epub 2013 May 23. PMID 23707554
- [Background] Cope EK, Lynch SV. Novel microbiome-based therapeutics for chronic rhinosinusitis. Curr Allergy Asthma Rep. 2015 Mar;15(3):504. doi: 10.1007/s11882-014-0504-y. PMID 25777787
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Lund VJ, Kennedy DW. Staging for rhinosinusitis. Otolaryngol Head Neck Surg. 1997 Sep;117(3 Pt 2):S35-40. doi: 10.1016/S0194-59989770005-6. PMID 9334786
- [Background] Greiff L, Andersson M, Persson CG. Nasal secretions and exudations : collection and approaches to analysis. Methods Mol Med. 2001;56:61-73. doi: 10.1385/1-59259-151-5:61. PMID 21336890
- [Background] Greiff L, Pipkorn U, Alkner U, Persson CG. The 'nasal pool' device applies controlled concentrations of solutes on human nasal airway mucosa and samples its surface exudations/secretions. Clin Exp Allergy. 1990 May;20(3):253-9. doi: 10.1111/j.1365-2222.1990.tb02680.x. PMID 2364306
- [Background] Morgan XC, Huttenhower C. Chapter 12: Human microbiome analysis. PLoS Comput Biol. 2012;8(12):e1002808. doi: 10.1371/journal.pcbi.1002808. Epub 2012 Dec 27. PMID 23300406
- [Background] Sahlstrand-Johnson P, Ohlsson B, Von Buchwald C, Jannert M, Ahlner-Elmqvist M. A multi-centre study on quality of life and absenteeism in patients with CRS referred for endoscopic surgery. Rhinology. 2011 Oct;49(4):420-8. doi: 10.4193/Rhino11.101. PMID 21991567